CLINICAL TRIAL: NCT02688309
Title: Pro-permeability and Pro-fibrosis Factors in the Aqueous of Patients With Retinal Diseases
Acronym: P3F2
Status: Terminated | Type: Observational
Why Stopped: Enrollment was affected due to the COVID-19 pandemic
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00045274
Record Dates: First submitted 2015-12-21; First posted 2016-02-23 (Estimated); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Macular Edema; Fibrosis of the Retina
MeSH Terms: conditions — Macular Edema | interventions — Calcium Dobesilate; Dexamethasone; Surgical Procedures, Operative; Paracentesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Clinic Patients: Patients from the clinic will be considered for enrollment if they are receiving an intraocular injection of a steroid as part of standard care for macular edema or progressive fibrosis.
  Clinic patients who are receiving an intraocular injection of steroid (Ozurdex) as part of standard care who agree to participate will have an anterior chamber (AC) tap just prior to the intraocular injection of steroid and a second AC tap at a follow up visit 6 ± 2 weeks after the steroid injection.
  Interventions: Drug: Ozurdex; Procedure: Anterior Chamber (AC) Tap
- OR Patients: Patients undergoing surgery for one of the following conditions: (1) Proliferative Diabetic Retinopathy, (2) rhegmatogenous retinal detachment with PVR, (3) rhegmatogenous retinal detachment without PVR, (4) macular pucker, (5) macular hole. Surgical patients who agree to participate will have an anterior chamber (AC) tap at the beginning of surgery.
  Interventions: Procedure: Surgery; Procedure: Anterior Chamber (AC) Tap

INTERVENTIONS:
Drug: Ozurdex — Patients from the clinic will be considered for enrollment if they are receiving an intraocular injection of a steroid as part of standard care for macular edema or progressive fibrosis. Clinic patients who are receiving an intraocular injection of steroid (Ozurdex) as part of standard care who agree to participate will have an AC tap just prior to the intraocular injection of steroid and a second AC tap at a follow up visit 6 ± 2 weeks after the steroid injection.
  Other Names: Dexamethasone intravitreal implant 0.7 mg
  Groups: Clinic Patients
Procedure: Surgery — The 60 patients from the operating room will be patients undergoing surgery for one of the following conditions: (1) Proliferative Diabetic Retinopathy, (2) rhegmatogenous retinal detachment with PVR, (3) rhegmatogenous retinal detachment without PVR, (4) macular pucker, (5) macula hole. All patients will be administered an AC (Anterior Chamber) tap just prior to the surgical procedure while in the OR.
  Groups: OR Patients
Procedure: Anterior Chamber (AC) Tap — A paracentesis removing about 0.1 ml of fluid from the front part of the eye (the aqueous chamber) will be performed in the operating room just prior to surgery or in the clinic. In the operating room, the AC tap is done after the eye is anesthetized and cleaned with 5% povidone iodine for the surgery. A 30-gauge needle attached to a tuberculin syringe is inserted into the AC and 0.1 ml of aqueous is removed. The wound is self-sealing and has no effect on the surgery. In the clinic, the AC tap is done after drops of proparacaine and 5% povidone iodine is placed in the eye and a lid speculum is inserted. The patient is seated at a slit lamp and a 30-gauge needle attached to a tuberculin syringe is inserted into the AC and 0.1 ml of aqueous is aspirated and then the needle is removed.

SUMMARY:
This study will examine potential factors in the aqueous humor that may contribute to the development or progression of macular edema or fibrosis (due to any underlying disease) in patients suffering from these conditions.

DETAILED DESCRIPTION:
The primary purpose of this study is to determine the correlation of pro-permeability and pro-fibrosis factor levels and downstream receptor/signaling molecule activation with disease activity in patients with macular edema or fibrosis secondary to any underlying disease.

120 patients will be enrolled from both the clinic and OR, with the latter patients undergoing surgery for proliferative diabetic retinopathy, rhegmatogenous retinal detachment with Proliferative vitreoretinopathy (PVR), rhegmatogenous retinal detachment without PVR, macular pucker, or macular hole. Clinic patients must be receiving an intraocular injection of a steroid as part of standard of care for macular edema or progressive fibrosis.

Surgical patients will receive an anterior chamber (AC) tap at the beginning of surgery, while clinic patients will receive an AC tap prior to the intraocular injection of steroid with a second AC tap at a follow-up visit 6 +/- 2 weeks after the first injection. The aqueous sample will then be analyzed by measuring the levels of various pro-permeability and pro-fibrosis factors and/or their downstream receptor/signaling molecule activation.

We will also determine the correlation between reductions in foveal thickness or improvements in visual acuity with changes in the aqueous levels of pro-permeability and pro-fibrosis factors from baseline to week 6 in the clinic group.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent and authorization of use and disclosure of protected health information
* Age >= 18 years
* Undergoing surgery as part of standard care for one of the following conditions: (1) Proliferative Diabetic Retinopathy (PDR), (2) rhegmatogenous retinal detachment with PVR, (3) rhegmatogenous retinal detachment without PVR, (4) macular pucker, (5) macular hole OR receiving as part of standard care, an intraocular injection of a steroid for macular edema or progressive fibrosis.

Exclusion Criteria:

* Previous use of an anti-Vascular Endothelial Growth Factor (VEGF) drug within 1 month of study entry
* Any condition that the investigator believes would pose a significant hazard to the subject if standard study procedures were conducted.
* Inability to comply with study or follow up procedures
* Patients with active or suspected ocular or periocular infection, including most viral diseases of the cornea and conjunctiva, including active epithelial herpes simplex keratitis (dendritic keratitis), vaccinia, varicella, mycobacterial infections, and fungal diseases.
* Pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Proliferative Diabetic Retinopathy, Rhegmatogeous Retinal detachment with and without PVR, Macular pucker, Macular hole, Macular Edema and Fibrosis of the Retina,
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2015-01-13 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Correlation of pro-permeability and pro-fibrosis factor levels and receptor/signaling molecule activation with disease activity. | Baseline

SECONDARY OUTCOMES:
Correlation between reduction in foveal thickness and changes in aqueous levels of pro-permeability and pro-fibrosis factors from baseline to week 6 in the clinic cohort. | Baseline, week 6.
Correlation between changes in visual acuity and changes in the aqueous levels of pro-permeability and pro-fibrosis factors from baseline to week 6 in the clinic cohort. | Baseline, week 6.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Campochiaro, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Wilmer Eye Institute, Baltimore, Maryland, United States

REFERENCES:
- [Background] Scholl S, Kirchhof J, Augustin AJ. Pathophysiology of macular edema. Ophthalmologica. 2010;224 Suppl 1:8-15. doi: 10.1159/000315155. Epub 2010 Aug 18. PMID 20714176
- [Background] Marmor MF. Mechanisms of fluid accumulation in retinal edema. Doc Ophthalmol. 1999;97(3-4):239-49. doi: 10.1023/a:1002192829817. PMID 10896337
- [Background] Tranos PG, Wickremasinghe SS, Stangos NT, Topouzis F, Tsinopoulos I, Pavesio CE. Macular edema. Surv Ophthalmol. 2004 Sep-Oct;49(5):470-90. doi: 10.1016/j.survophthal.2004.06.002. PMID 15325193
- [Background] Aiello LP, Avery RL, Arrigg PG, Keyt BA, Jampel HD, Shah ST, Pasquale LR, Thieme H, Iwamoto MA, Park JE, et al. Vascular endothelial growth factor in ocular fluid of patients with diabetic retinopathy and other retinal disorders. N Engl J Med. 1994 Dec 1;331(22):1480-7. doi: 10.1056/NEJM199412013312203. PMID 7526212
- [Background] Vinores SA, Youssri AI, Luna JD, Chen YS, Bhargave S, Vinores MA, Schoenfeld CL, Peng B, Chan CC, LaRochelle W, Green WR, Campochiaro PA. Upregulation of vascular endothelial growth factor in ischemic and non-ischemic human and experimental retinal disease. Histol Histopathol. 1997 Jan;12(1):99-109. PMID 9046048
- [Background] Lima e Silva R, Shen J, Hackett SF, Kachi S, Akiyama H, Kiuchi K, Yokoi K, Hatara MC, Lauer T, Aslam S, Gong YY, Xiao WH, Khu NH, Thut C, Campochiaro PA. The SDF-1/CXCR4 ligand/receptor pair is an important contributor to several types of ocular neovascularization. FASEB J. 2007 Oct;21(12):3219-30. doi: 10.1096/fj.06-7359com. Epub 2007 May 23. PMID 17522382
- [Background] Oshima Y, Deering T, Oshima S, Nambu H, Reddy PS, Kaleko M, Connelly S, Hackett SF, Campochiaro PA. Angiopoietin-2 enhances retinal vessel sensitivity to vascular endothelial growth factor. J Cell Physiol. 2004 Jun;199(3):412-7. doi: 10.1002/jcp.10442. PMID 15095288
- [Background] Campochiaro PA, Hafiz G, Channa R, Shah SM, Nguyen QD, Ying H, Do DV, Zimmer-Galler I, Solomon SD, Sung JU, Syed B. Antagonism of vascular endothelial growth factor for macular edema caused by retinal vein occlusions: two-year outcomes. Ophthalmology. 2010 Dec;117(12):2387-2394.e1-5. doi: 10.1016/j.ophtha.2010.03.060. Epub 2010 Jul 13. PMID 20630595